CLINICAL TRIAL: NCT03284840
Title: NUTRIHEALTH - Adults Nutrition as a Protective or Health-risk Factor
Brief Title: Adults Nutrition as a Protective or Health-risk Factor
Acronym: NUTRIHEALTH
Status: Completed | Type: Observational
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: National Institute of Public Health, Slovenia (Other Government); University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: KME72/07/16
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-02

CONDITIONS: Nutritional Status; Nutrient Deficiency; Micronutrient Deficiency; Vitamin D Deficiency; Vitamin B 12 Deficiency; Folic Acid Deficiency; Iron-deficiency; Thyroid Diseases; Diet
Keywords: dietary intake; nutritional status; micronutrients; thyroid health
MeSH Terms: conditions — Vitamin D Deficiency; Vitamin B 12 Deficiency; Folic Acid Deficiency; Anemia, Iron-Deficiency; Thyroid Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be freezed for possible further analyses on markers related with nutrition & health
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults (18-65 years)
  Interventions: Diagnostic Test: Assessement of nutritional status; Diagnostic Test: Thyroid size
- Elderly (65-74 years)
  Interventions: Diagnostic Test: Assessement of nutritional status; Diagnostic Test: Thyroid size

INTERVENTIONS:
Diagnostic Test: Assessement of nutritional status — Nutritional status for vitamin D, folic acid, vitamin B12 and iron.
Diagnostic Test: Thyroid size — Thyroid size by ultrasound.

SUMMARY:
To obtain up-to-date data on nutrient intakes in adults, a national dietary survey - the EU Menu study will be conducted during 12 consecutive months in 2017/2018, providing data on the consumption of foods and enabling the assessment of energy and macronutrient intakes. Participating subjects will be invited to NUTRIHEALTH study for assessment for micronutrient status (focusing into vitamin D, folic acid, vitamin B12, and iron) and medical examination, in which thyroid size will be aslo measured, to investigated thyroid epidemiology in Slovenia.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Republic of Slovenia (included to the register of residents)
* Finished EU MENU Slovenia Study

Exclusion Criteria:

* Not willing to give blood&urine sample
* Long-term disease
* Living in institutions with controled diet, such as such as in elderly care, hospital, prison, etc.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This observational study is conducted on randomly selected residents of Republic of Slovenia. The EU Menu study (LOT2) include a minimum of 1.133 of habitants from Slovenia in the age 18-74 years. In line with the EU Menu methodology and to ensure representativeness of the sample, participants will be randomly selected from the Slovenian population using Central Population Register (selection outsourced by the Statistical Office of Republic of Slovenia ), and visited on their home. After completion of the EU Menu Survey (questionnaires on self-reported health status and food intake), participants will be invited to collaborate in the proposed study.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of inadequate vitamin D status | 1 year
  epidemiology of vitamin D status will be investigated
Assessment of thyroid health | 1 year
  epidemiology of thyroid Health will be investigated

SECONDARY OUTCOMES:
Assessment of inadequate vitamin B12 status | 1 years
  epidemiology of vitamin 12 status will be investigated
Assessment of inadequate folic acid status | 1 years
  epidemiology of folic acid status will be investigated
Assessment of inadequate iron status | 1 years
  epidemiology of iron status will be investigated

CONTACTS AND LOCATIONS:
Overall Officials: Igor Pravst, PhD, Study Chair — Nutrition Institute, Ljubljana
Locations (3):
- Slovenia (3):
  - National Institute of Public Health, Slovenia, Ljubljana
  - Nutrition Institute, Ljubljana, Ljubljana
  - University Medical Centre Ljubljana, Ljubljana